CLINICAL TRIAL: NCT03478644
Title: Clinical Study To Determine The Oral and Dermal Tolerability of an Experimental Denture Wipe
Brief Title: Oral and Dermal Tolerability Clinical Study of an Experimental Denture Wipe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 203115
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2018-08-31 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-07

CONDITIONS: Denture Cleansers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The dental examiner and dermatologist blinded for both treatment arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental Denture Wipe (Experimental): Participants of this arm were instructed to use the experimental wipe to clean their dentures up to 4 times daily.
  Interventions: Device: Experimental Denture Wipe
- Tap Water (Placebo Comparator): Participants of this arm were instructed to use running tap water to clean their dentures up to 4 times daily.
  Interventions: Other: Tap Water

INTERVENTIONS:
Device: Experimental Denture Wipe — Participants were instructed to use the experimental wipe to clean their dentures, external to their mouth, up to 4 times daily (once after completion of each of their three main meals and once at any other time) for 14 days. Participants were instructed to use one wipe per denture.
  Arms: Experimental Denture Wipe
Other: Tap Water — Participants were instructed to use running tap water to clean their dentures up to 4 times daily (once after completion of each of their three main meals and once at any other time) for 14 days.
  Arms: Tap Water

SUMMARY:
The purpose of this two-phase study was to evaluate the oral and dermal tolerance of an experimental, non-rinse denture cleansing wipe after 7 and 14 days of use. In addition, the consumer acceptability of the denture cleansing wipes was also evaluated via a consumer acceptability questionnaire. A methodology was also evaluated to assess the efficacy of the denture wipe at removing food debris as exploratory objective.

DETAILED DESCRIPTION:
This was a two phase single-center study. Phase 1 (Food removal testing), was monadic and only the wipe treatment was administered to complete upper dentures. Phase 1 participants then progressed to phase 2 (oral soft tissue [OST] and dermal assessment) which was an examiner blind parallel group, randomized and stratified (by denture type) design where both treatments (a single wipe and water control) were administered. Phase 2 participants included both fully and partially edentulous adult participants. Participants were not permitted to use any denture cleansers other than those provided and were not permitted to use denture fixatives for the duration of the study. The study comprised a Screening/Baseline visit and a 2 week Treatment Period with visits after 1 and 2 weeks use. Following screening participants who were eligible for Phase 1 were assessed for food migration adequacy. Participants consumed 30-32g (gram) of non-salted peanut halves in a controlled manner, then briefly rinsed their mouth with water and removed their upper denture. The investigator visually assessed the peanut particle migration underneath the denture on a 0-3 scale and those participants with a score greater than 0 were wiped by the participant with the experimental denture wipe. The mass of peanuts removed by the wipe and those remaining on the denture was subsequently measured. For a subset of participants (2 participants per peanut particle migration scale score), their dentures were photographed after peanut consumption both before and after use of the experimental denture wipe. Phase 1 participants then continued into Phase 2. All Phase 2 participants undertook an OST examination and a dermatological assessment of both sides of their lead hand, then randomized. The dental examiner and dermatologist were blinded to the treatment allocation. The results of these assessments served as the baseline reading. Participants were then instructed on the use of their assigned treatment with the first application undertaken and supervised at the study site. Participants were provided with a diary card to record their treatment applications and a consumer acceptability questionnaire to be completed at the time of their first at home treatment use. Participants were also provided with denture cleansing tablets for use overnight for the duration of the study in order to maintain denture hygiene. Participants returned to the study site after 7±3 and 14±3 days use of product for repeat OST and dermatological assessments.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated understanding of the study procedures, restrictions and was willing to participate as evidenced by voluntary written informed consent and had received a signed and dated copy of the informed consent form.
* Understood and was willing, able and comply with all study procedures and restrictions.
* Participant was in good general and mental health with, in the opinion of the investigator or medically qualified designee - (a) no clinically significant and relevant abnormalities of medical or physical history; (b) absence of any condition that impacted on the participant's safety or well-being or affected the individual's ability to understand and follow study procedures.
* Denture Requirements, fully or partially edentulous: (a) Phase 1 eligible participants had a full upper denture and may Have a full or partial lower denture or no lower Denture; (b) Phase 2 eligible subjects will have at least one full or partial denture; (c) Dentures considered in good condition according to the investigator or dental examiner, with no damage according to assessment criteria; (d) Participants with a peanut particle migration rating greater than zero on the upper denture only for participants screened for food removal testing.
* Skin Phototype (Fitzpatrick), I to IV, according to the scale only skin phototypes I to IV are acceptable for inclusion in this study: Type I - White; very fair; freckles; typical albino skin. Always burns, never tans, Type II -White; fair. Usually burns, tans with difficulty, Type III - Beige; very common. Sometimes mild burn, gradually tans to a light brown, Type IV - Beige with a brown tint; typical Mediterranean Caucasian skin. Rarely burns, tans with ease to a moderate brown, Type V - Dark brown. Very rarely burns, tans very easily, Type VI Black - Never burns, tans very easily, deeply pigmented.

Exclusion Criteria:

* Women who were known to be pregnant or who were intending to become pregnant over the duration of the study.
* Women who were breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients. Known allergy to any nuts or peanuts. History of allergic reactions or intense feelings of discomfort to topically used products: cosmetics or drugs.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit, except for participants who were enrolled on GSKCH study 205915 who might enrolled onto this study 7 days after their completion of 205915. Previous participation in this study.
* Recent history (within the last one year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Denture adhesive users were excluded from this study.
* Participants with OST findings such as, stomatitis, open sores, lesions, redness or swelling were excluded.
* Other Conditions because of participants were excluded are as follows: History of swallowing or choking difficulties; participants unwilling to refrain from using their existing denture cleansing routine for the duration of the study; taking or have taken a bisphosphonate drug for treatment of osteoporosis; skin marks in the experimental area which may interfere with the evaluation of potential skin reactions; active skin diseases (local and/or disseminated) that may interfere with the study results; participants with immunodeficiencies, intense sunlight exposure or tanning session within 15 days before the baseline evaluation or during the study that has resulted in sunburn; body cosmetic and/or dermatological treatment until three weeks before screening or during the study; continual use of therapeutic, topical or systemic use of the following drugs: immunosuppressants, antihistamines, non-steroidal anti-inflammatory drugs and corticosteroids within two weeks before the screening for chronic conditions; oral or topical treatment with vitamin A acid and/or its derivatives within one month before start of study; vaccination within three weeks before or during the study; participants with dermographism; any condition not previously mentioned that in the investigator's opinion may impair the study evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at one center in the United States.
Pre-assignment Details: A total of 155 participants were screened, of which first 31 eligible participants with complete upper dentures were included in Phase 1 (food removal testing). Out of 155 participants, 152 were randomized in Phase 2 (oral soft tissue and dermal assessment). 3 participants were not randomized as 2 were screened failure and 1 withdrew from study.
Groups:
- Experimental Denture Wipe: All the participants of this arm were instructed to use the experimental wipe to clean their dentures up to 4 times daily.
- Water Rinse: All the participants of this arm were instructed to use running tap water to clean their dentures up to 4 times daily.
Period: Phase 1
Arm/Group | Experimental Denture Wipe | Water Rinse
Started | 31 (In Phase 1, only the wipe treatment was administered to eligible participants.) | 0
Completed | 31 (In Phase 1, only the wipe treatment was administered to eligible participants.) | 0
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Experimental Denture Wipe | Water Rinse
Started | 76 | 76
Completed | 73 | 75
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline assessment was performed on safety population, which included all participants who were randomized and received treatment at least once during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Denture Wipe | Water Rinse | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.99 (12.702) | 61.03 (12.622) | 61.01 (12.620)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 48 | 105
  Male | 19 | 28 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 8 | 18
  White | 64 | 67 | 131
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Experiencing or Reporting Treatment Emergent (TE) Oral Adverse Events (AEs) on or Before 14 Days of Use
Description: Proportion of participants experiencing or reporting TE oral AEs on or before 14 days of use treatments were reported. TE AEs include AEs that were identified during an oral soft tissue examination, a dermal assessment or reported by the subject. AEs were categorized as oral or non-oral by the Clinical Research scientist prior to database lock (oral AE's were AEs effecting tissues associated with the oral cavity extending from the labial mucosa to the pharyngeal area).
Time Frame: up to 14 days
Population: Analysis for this outcome was performed on safety population which included all the participants who were randomized and received treatment at least once during the study. No inferential statistical analysis has been performed for this outcome.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Water Rinse: Participants of this arm were instructed to use running tap water to clean their dentures up to 4 times daily.
Arm/Group | Experimental Denture Wipe | Water Rinse
Number analyzed (Participants) | 76 | 76
Proportion of participants | 0.039 [0.01 to 0.11] | 0.013 [0.00 to 0.07]

2. Primary Outcome: Proportion of Participants Experiencing or Reporting Treatment Emergent (TE) Oral Adverse Events (AEs) on or Before 7 Days of Use
Description: Proportion of participants experiencing or reporting TE oral AEs on or before 7 days of use treatments were reported. TE AEs include AEs that were identified during an oral soft tissue examination, a dermal assessment or reported by the subject. AEs were categorized as oral or non-oral by the Clinical Research scientist prior to database lock (oral AE's were AEs effecting tissues associated with the oral cavity extending from the labial mucosa to the pharyngeal area).
Time Frame: up to 7 days
Population: Analysis for this outcome was performed on safety population which included all participants who were randomized and received treatment at least once during the study. No inferential statistical analysis has been performed for this outcome.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Experimental Denture Wipe | Water Rinse
Number analyzed (Participants) | 76 | 76
Proportion of participants | 0.013 [0.00 to 0.07] | 0.000 [0.00 to 0.05]

3. Secondary Outcome: Proportion of Participants Experiencing Skin Irritation Scores of 2 or Greater After 7 and 14 Days of Use
Description: Dermal assessment performed by a suitably qualified dermatologist on the front and back of the participant's dominant hand (hand with which participant used to hold the wipe during use) using skin irritation score that range from 0-4 as follows: 0 = no apparent cutaneous involvement, 0.5= equivocal reaction, 1= slight erythema with or without oedema, 2= moderate erythema, oedema with or without papules, 3= severe erythema, oedema with or without papules, 4= severe erythema, oedema with vesicles or blisters. Any site where skin irritation was scored ≥2, was visually assessed and reported.
Time Frame: Day 7, Day 14
Population: Analysis for this outcome was performed on safety population which included all participants who were randomized and received treatment at least once during the study.
Measure: Number; unit: Proportion of participants
Arm/Group | Experimental Denture Wipe | Water Rinse
Number analyzed (Participants) | 76 | 76
Proportion of participants
  At Day 7 | 0 | 0
  At Day 14 | 0 | 0

4. Secondary Outcome: Number of Participants Responses for Consumer Acceptability Questionnaire Score
Description: All the participants supplied with a consumer acceptability questionnaire (Question [Q] 1 to 4) to complete immediately before & after their first use of treatment at home after eating a meal. The number of participants with individual score was reported. After eating & before cleaning denture: Q1= how fresh does denture feel?, Q2= how clean does denture feel?; Look in the mirror and smile, now answer the following questions: Q3= after eating & before cleaning, how clean does denture/smile look ?, Q4= after removing & cleaning denture, how fresh does denture feel?, Q5= after removing & cleaning denture, run your tongue over denture teeth, how clean does denture feel?, Q6= after removing & cleaning denture, how clean does denture/smile look?, Q7= after removing & cleaning denture, how satisfied are you with amount of debris removed? All questions were scored as follows for respective parameter(fresh/clean/satisfied): 0=Not at all, 1=slightly, 2=moderately, 3=very, 4=extremely.
Time Frame: Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Denture Wipe | Water Rinse
Number analyzed (Participants) | 76 | 76
Participants
  Q1: Score 0 - Not fresh at all | 20 | 18
  Q1: Score 1 - Slightly fresh | 16 | 26
  Q1: Score 2 - Moderately fresh | 18 | 17
  Q1: Score 3 - Very fresh | 14 | 10
  Q1: Score 4 - Extremely fresh | 8 | 5
  Q2: Score 0 - Not clean at all | 12 | 12
  Q2: Score 1 - Slightly clean | 12 | 23
  Q2: Score 2 - Moderately clean | 26 | 21
  Q2: Score 3 - Very clean | 15 | 14
  Q2: Score 4 - Extremely clean | 11 | 6
  Q3: Score 0 - Not clean at all | 5 | 1
  Q3: Score 1 - Slightly clean | 15 | 15
  Q3: Score 2 - Moderately clean | 23 | 31
  Q3: Score 3 - Very clean | 23 | 21
  Q3: Score 4 - Extremely clean | 10 | 8
  Q4: Score 0 - Not fresh at all | 0 | 0
  Q4: Score 1 - Slightly fresh | 0 | 3
  Q4: Score 2 - Moderately fresh | 11 | 22
  Q4: Score 3 - Very fresh | 32 | 31
  Q4: Score 4 - Extremely fresh | 33 | 20
  Q5: Score 0 - Not clean at all | 0 | 1
  Q5: Score 1 - Slightly clean | 1 | 0
  Q5: Score 2 - Moderately clean | 9 | 18
  Q5: Score 3 - Very clean | 32 | 37
  Q5: Score 4 - Extremely clean | 34 | 20
  Q6: Score 0 - Not clean at all | 0 | 0
  Q6: Score 1 - Slightly clean | 1 | 1
  Q6: Score 2 - Moderately clean | 10 | 18
  Q6: Score 3 - Very clean | 33 | 37
  Q6: Score 4 - Extremely clean | 32 | 20
  Q7: Score 0 - Not satisfied at all | 0 | 0
  Q7: Score 1 - Slightly satisfied | 0 | 0
  Q7: Score 2 - Moderately satisfied | 9 | 21
  Q7: Score 3 - Very satisfied | 40 | 36
  Q7: Score 4 - Extremely satisfied | 27 | 19

ADVERSE EVENTS:
Time Frame: Approximately 17 days (from Screening Visit to Visit 3)
Arm/Group | Experimental Denture Wipe | Water Rinse
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 3/76 | 1/76
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Denture Wipe (N=76) | Water Rinse (N=76)
Mouth Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lip Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.